CLINICAL TRIAL: NCT01052545
Title: Guideline Implementation to Decrease Inappropriate Bacteriuria Treatment
Brief Title: Asymptomatic Bacteriuria Guideline Implementation Study
Acronym: ABU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 09-104; H-24180 (Other Grant/Funding Number: HSR&D Service)
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Infection Due to Indwelling Urinary Catheter; Asymptomatic Bacteriuria
Keywords: urinary tract infection; urinary catheter; bacteriuria; clinical guidelines; audit-feedback; guidelines implementation
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1- Intervention: Audit-Feedback (Experimental): Baseline surveillance for the clinical outcomes will begin in year 1 at the intervention site and continue for all 3 years of the project. Guideline distribution will begin in year 2 and continue throughout the project. Audit-feedback will occur during year 2 of the study at the intervention site. Feedback will be delivered to individual health care providers at the intervention site during year 2.Unit-level audit feedback will be delivered at the intervention site during years 2 and 3 of the study. Provider surveys of knowledge and attitudes concerning the ABU guidelines will be administered at the intervention site in years 2 and 3 of the project.
  Interventions: Behavioral: Audit-Feedback
- Arm 2- Control (No Intervention): At the control site, baseline surveillance for the clinical outcomes will begin in year 1 at the and continue for all 3 years of the project. Guideline distribution will begin in year 2 and continue throughout the project. Audit-feedback will not occur at the control site. Provider surveys of knowledge and attitudes concerning the ABU guidelines will be administered at the control site in year 3 of the project.

INTERVENTIONS:
Behavioral: Audit-Feedback — Applied as a post-prescription antimicrobial review based on established guidelines.
  Arms: Arm 1- Intervention: Audit-Feedback

SUMMARY:
Overtreatment of asymptomatic bacteriuria (ABU) is a quality, safety, and cost issue, particularly as unnecessary antibiotics lead to emergence of resistant pathogens. The investigators' proposal to bring clinical practice in line with published guidelines has significant potential to reduce unnecessary antibiotic use for ABU in the VA healthcare system, thus improving the quality and safety of veterans' healthcare. The investigators' study will also provide important insights about how to implement and sustain evidence-based clinical practice within VA hospitals.

DETAILED DESCRIPTION:
Anticipated Impacts on Veterans' Healthcare: Urinary tract infection (UTI) is the single most common hospital-acquired infection. However, the majority of cases of nosocomial catheter-associated urinary tract infection (CAUTI) are really asymptomatic bacteriuria (ABU). ABU is not a clinically significant condition, and treatment is unlikely to confer benefit. Overtreatment of ABU is a quality, safety, and cost issue, particularly as unnecessary antibiotics lead to emergence of resistant flora. The proposal to bring clinical practice in line with published guidelines has significant potential to decrease CAUTI and associated inappropriate antibiotic use in VA hospitals. The study will also provide information about how to maximize effectiveness of audit-feedback to achieve guideline adherence in the inpatient VA setting.

Project Background/Rationale: Evidence-based guidelines recommend that providers neither screen for nor treat ABU in most catheterized patients. However, a significant gap between these guidelines and clinical practice has been documented at the investigators' VA hospital and throughout the world. Since many VA patients in both acute care settings and sub-acute care settings, such as intermediate and long-term care, have a legitimate need for a urinary catheter, the issue of overtreatment of catheter-associated ABU is an active problem for the VA.

Project Objectives: The investigators hypothesize that implementing the existing evidence-based guidelines about non-treatment of ABU will dramatically reduce the unnecessary use of antibiotics to treat ABU and the incidence of incorrectly diagnosed CAUTI. The first objective is to improve quality of care concerning ABU in terms of specific clinical outcomes (inappropriate screening for and treatment of ABU) through implementation of an audit-feedback strategy. The investigators also hypothesize that successful implementation of an audit-feedback strategy will result in measurable changes in clinicians' knowledge and attitudes concerning ABU practice guidelines. The second objective is to assess through surveys the effect of the implementation on clinicians' guideline awareness, familiarity, acceptance, and outcome expectancy.

Project Methods: The investigators' guidelines implementation strategy will employ audit-feedback, applied as a post-prescription antimicrobial review based on established guidelines. The study population for the clinical outcomes is all inpatients on certain wards at the intervention site (Houston VA) and the control site (San Antonio VA). The investigators' study population for the audit-feedback intervention and surveys is the health care providers on these wards. The investigators propose a 3-year study. During the first year the investigators will observe the baseline incidence of inappropriate screening for and treatment of ABU at both sites. Blinded monitoring of clinical outcomes will continue during the next 2 years of the study. During the second year, the investigators will distribute the guidelines at both sites. Clinicians at the intervention site will receive individualized feedback, either by telephone or in person, about whether their management of bacteriuria was guideline-compliant. Unit-level feedback will also be provided. During the third year, individualized feedback will cease, but unit-level feedback will continue as this constitutes a sustainable intervention. Clinicians will complete pre/post surveys of awareness, familiarity, acceptance, and outcome expectancy at the intervention site in year 2 and at both sites in year 3. Differences in outcomes between the individualized intervention in year 2 and the group-level intervention in year 3 will help to determine the necessary intensity of intervention for dissemination and implementation in other VA facilities.

ELIGIBILITY:
Inclusion Criteria:

* For Objective 1 (Clinical Outcomes), all inpatients at the MEDVAMC or STVHCS on the units of interest (medicine or ECL) during the 3 year period of the study will be included in the chart review process.
* For Objective 2, modifying health care provider knowledge and behavior through audit-feedback and surveys, the investigators will attempt to involve all health care providers on rotation at the VA on the targeted wards during the study period.
* The audit-feedback intervention will be applied to the health care providers on the targeted wards who make the decision to treat CAUTI.

Exclusion Criteria:

* None.
* For the chart review component, the investigators want to capture all available data about the clinical outcomes during the study period.

  * review the inpatient rosters on the wards of interest several times per week to determine how many of the patients have urinary catheters, etc.
  * survey as many health care providers as possible who rotate on the wards of interest during the study period.
  * the investigators anticipate that all health care providers who work at the VA hospital will be competent to provide or refuse consent to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1598 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Trautner, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

REFERENCES:
- [Background] Lin E, Bhusal Y, Horwitz D, Shelburne SA 3rd, Trautner BW. Overtreatment of enterococcal bacteriuria. Arch Intern Med. 2012 Jan 9;172(1):33-8. doi: 10.1001/archinternmed.2011.565. PMID 22232145
- [Background] Trautner BW. Asymptomatic bacteriuria: when the treatment is worse than the disease. Nat Rev Urol. 2011 Dec 6;9(2):85-93. doi: 10.1038/nrurol.2011.192. PMID 22143416
- [Background] Gupta K, Trautner BW. Diagnosis and management of recurrent urinary tract infections in non-pregnant women. BMJ. 2013 May 29;346:f3140. doi: 10.1136/bmj.f3140. No abstract available. PMID 23719637
- [Background] Trautner BW. Management of catheter-associated urinary tract infection. Curr Opin Infect Dis. 2010 Feb;23(1):76-82. doi: 10.1097/QCO.0b013e328334dda8. PMID 19926986
- [Result] Burns AC, Petersen NJ, Garza A, Arya M, Patterson JE, Naik AD, Trautner BW. Accuracy of a urinary catheter surveillance protocol. Am J Infect Control. 2012 Feb;40(1):55-8. doi: 10.1016/j.ajic.2011.04.006. Epub 2011 Aug 3. PMID 21813209
- [Result] Trautner BW, Kelly PA, Petersen N, Hysong S, Kell H, Liao KS, Patterson JE, Naik AD. A hospital-site controlled intervention using audit and feedback to implement guidelines concerning inappropriate treatment of catheter-associated asymptomatic bacteriuria. Implement Sci. 2011 Apr 22;6:41. doi: 10.1186/1748-5908-6-41. PMID 21513539
- [Result] Trautner BW, Patterson JE, Petersen NJ, Hysong S, Horwitz D, Chen GJ, Grota P, Naik AD. Quality gaps in documenting urinary catheter use and infectious outcomes. Infect Control Hosp Epidemiol. 2013 Aug;34(8):793-9. doi: 10.1086/671267. Epub 2013 Jun 17. PMID 23838219
- [Result] Kizilbash QF, Petersen NJ, Chen GJ, Naik AD, Trautner BW. Bacteremia and mortality with urinary catheter-associated bacteriuria. Infect Control Hosp Epidemiol. 2013 Nov;34(11):1153-9. doi: 10.1086/673456. Epub 2013 Sep 23. PMID 24113598
- [Result] Trautner BW, Bhimani RD, Amspoker AB, Hysong SJ, Garza A, Kelly PA, Payne VL, Naik AD. Development and validation of an algorithm to recalibrate mental models and reduce diagnostic errors associated with catheter-associated bacteriuria. BMC Med Inform Decis Mak. 2013 Apr 15;13:48. doi: 10.1186/1472-6947-13-48. PMID 23587259
- [Result] Grigoryan L, Abers MS, Kizilbash QF, Petersen NJ, Trautner BW. A comparison of the microbiologic profile of indwelling versus external urinary catheters. Am J Infect Control. 2014 Jun;42(6):682-4. doi: 10.1016/j.ajic.2014.02.028. PMID 24837121
- [Result] Trautner BW, Grigoryan L. Approach to a positive urine culture in a patient without urinary symptoms. Infect Dis Clin North Am. 2014 Mar;28(1):15-31. doi: 10.1016/j.idc.2013.09.005. Epub 2013 Dec 8. PMID 24484572
- [Result] Trautner BW, Grigoryan L, Petersen NJ, Hysong S, Cadena J, Patterson JE, Naik AD. Effectiveness of an Antimicrobial Stewardship Approach for Urinary Catheter-Associated Asymptomatic Bacteriuria. JAMA Intern Med. 2015 Jul;175(7):1120-7. doi: 10.1001/jamainternmed.2015.1878. PMID 26010222
- [Result] Grigoryan L, Naik AD, Horwitz D, Cadena J, Patterson JE, Zoorob R, Trautner BW. Survey finds improvement in cognitive biases that drive overtreatment of asymptomatic bacteriuria after a successful antimicrobial stewardship intervention. Am J Infect Control. 2016 Dec 1;44(12):1544-1548. doi: 10.1016/j.ajic.2016.04.238. Epub 2016 Jul 7. PMID 27397910
- [Result] Naik AD, Skelton F, Amspoker AB, Glasgow RA, Trautner BW. A fast and frugal algorithm to strengthen diagnosis and treatment decisions for catheter-associated bacteriuria. PLoS One. 2017 Mar 28;12(3):e0174415. doi: 10.1371/journal.pone.0174415. eCollection 2017. PMID 28350833
- [Derived] Hysong SJ, Kell HJ, Petersen LA, Campbell BA, Trautner BW. Theory-based and evidence-based design of audit and feedback programmes: examples from two clinical intervention studies. BMJ Qual Saf. 2017 Apr;26(4):323-334. doi: 10.1136/bmjqs-2015-004796. Epub 2016 Jun 10. PMID 27288054

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The investigators reviewed the electronic medical record continuously at both sites to detect urine cultures and antibiotic use. At the intervention site, we reviewed 170,345 bed days over the 3 years of the project, while at the control site, we reviewed 119,409 bed days over the same time period. The intervention was delivered to the providers.
Pre-assignment Details: From the bed days reviewed, we determined which patient had a positive urine culture that was associated with the presence of a urinary catheter. These cases were studied further to determine if antimicrobial use was compliant with guidelines or non-compliant. These cases became the numbers "enrolled" in each arm of this study.
Groups:
- Arm 1- Intervention: Audit-Feedback: Year 1: baseline surveillance at both sites Year 2: case based, individual audit and feedback delivered to providers, a guidelines based diagnostic algorithm for CAUTI versus asymptomatic bacteriuria (ASB) was given to providers and reinforced in the audit and feedback sessions.
  Year 3: cased based, group audit and feedback delivered to providers, again based on this diagnostic algorithm.
  Audit-Feedback: Applied as a post-prescription antimicrobial review based on established guidelines.
- Arm 2- Control: This was the contemporary control group. Surveillance for the outcomes of interest (urine cultures order and antibiotics used to treat urine cultures) continued for all 3 years. Providers at this site received standard education about the CAUTI and asymptomatic bacteriuria guidelines delivered in a grand rounds format, and they also received a PDF of the full guidelines by email.
Period: Overall Study
Arm/Group | Arm 1- Intervention: Audit-Feedback | Arm 2- Control
Started | 867 | 731
Completed | 867 | 731
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1-Intervention: Audit-Feedback: Baseline surveillance for the clinical outcomes will begin in year 1 at the intervention site and continue for all 3 years of the project. Guideline distribution will begin in year 2 and continue throughout the project. Audit-feedback will occur during year 2 of the study at the intervention site. Feedback will be delivered to individual health care providers at the intervention site during year 2.Unit-level audit feedback will be delivered at the intervention site during years 2 and 3 of the study. Provider surveys of knowledge and attitudes concerning the ABU guidelines will be administered at the intervention site in years 2 and 3 of the project.
  Audit-Feedback: Applied as a post-prescription antimicrobial review based on established guidelines.
- Total: Total of all reporting groups
Arm/Group | Arm 1-Intervention: Audit-Feedback | Arm 2- Control | Total
Number analyzed (Participants) | 867 | 731 | 1598
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (12) | 72 (13) | 72 (12)
Sex/Gender, Customized [Number; unit: participants] — *data missing for 43 pts
  participants
    Female | 19 | 19 | 38
    Male | 816 | 701 | 1517
Urinary catheter type [Number; unit: participants] — *data missing for 2 pts
  participants
    Foley | 510 | 444 | 954
    Condom | 341 | 160 | 501
    other | 15 | 126 | 141
Department [Number; unit: participants] — *data missing for 5 pts
  participants
    Medicine | 609 | 594 | 1203
    Longterm Care | 258 | 132 | 390

OUTCOME MEASURES:

1. Primary Outcome: Number of Cases of ABU That Are Treated Inappropriately With Antibiotics
Time Frame: Years 1, 2, & 3
Measure: Number (95% Confidence Interval); unit: cases/1,000 bed-days
Arm/Group | Arm 1-Intervention: Audit-Feedback | Arm 2- Control
Number analyzed (Participants) | 180 | 65
cases/1,000 bed-days
  Year 1 ASB tx | 1.6 [1.2 to 1.8] | 0.6 [0.3 to 0.9]
  Year 2 ASB tx | 0.5 [0.3 to 0.8] | 0.6 [0.3 to 0.6]
  Year 3 ASB tx | 0.4 [0.1 to 0.6] | 0.5 [0.3 to 0.7]

2. Primary Outcome: Urine Cultures Ordered
Description: Number of urine cultures collected per 1000 catheter-days for each unit
Time Frame: three years
Population: For this outcome measure, the number of participants is the number of patients that had urine cultures ordered. One patient could have multiple cultures ordered. Arm 1=5209 urine cultures ordered. Arm 2=5979 urine cultures ordered. This number was standardized by bed-days. Arm 1=170345 bed-days. Arm 2=119409 bed-days.
Measure: Number (95% Confidence Interval); unit: Total ucx ordered/1,000 bed-days
Groups:
- Intervention Group: Medicine and extended care wards at the intervention site
- Control Group: Medicine and extended care wards at control site
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 867 | 731
Total ucx ordered/1,000 bed-days
  Year 1 | 41.2 [37.0 to 45.3] | 49.3 [46.0 to 52.6]
  Year 2 | 23.3 [17.5 to 28.9] | 54.4 [51.4 to 57.5]
  Year 3 | 12.0 [8.8 to 15.1] | 46.6 [44.0 to 49.2]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.05, Regression, Logistic — Descriptive statistics were used to estimate the incidence rates per 1,000 bed-days and 95% confidence intervals (CI) for urine cultures ordered, ASB overtreatment and CAUTI under-treatment in each study period; to test whether there was a significant difference in monthly urine cultures ordered between the two study sites over time

3. Primary Outcome: Number of Cases of CAUTI Inappropriately Under-treated (no Antibiotics Given)
Time Frame: Years 1, 2, & 3
Measure: Number (95% Confidence Interval); unit: cases/1,000 bed-days
Arm/Group | Arm 1-Intervention: Audit-Feedback | Arm 2- Control
Number analyzed (Participants) | 27 | 17
cases/1,000 bed-days
  Year 1 CAUTI not tx | 0.2 [0.1 to 0.3] | 0.1 [0 to 0.3]
  Year 2 CAUTI not tx | 0.1 [0.02 to 0.3] | 0.2 [0.02 to 0.4]
  Year 3 CAUTI not tx | 0.05 [0 to 0.13] | 0.07 [0 to 0.1]

4. Secondary Outcome: Number of Days Antibiotics Are Given to Treat ABU
Time Frame: one year
Population: This data was not collected and is therefore not available.
Groups:
- Arm 1: Baseline surveillance for the clinical outcomes will begin in year 1 at the intervention site and continue for all 3 years of the project. Guideline distribution will begin in year 2 and continue throughout the project. Audit-feedback will occur during year 2 of the study at the intervention site. Feedback will be delivered to individual health care providers at the intervention site during year 2.Unit-level audit feedback will be delivered at the intervention site during years 2 and 3 of the study. Provider surveys of knowledge and attitudes concerning the ABU guidelines will be administered at the intervention site in years 2 and 3 of the project.
  Audit-Feedback: Applied as a post-prescription antimicrobial review based on established guidelines.
- Arm 2: At the control site, baseline surveillance for the clinical outcomes will begin in year 1 at the and continue for all 3 years of the project. Guideline distribution will begin in year 2 and continue throughout the project. Audit-feedback will not occur at the control site. Provider surveys of knowledge and attitudes concerning the ABU guidelines will be administered at the control site in year 3 of the project.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Clinicians' Awareness of and Familiarity With the ABU Guidelines.
Time Frame: one year
Population: health care practitioners
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Intervention Group; Post-intervention Group: Medicine and extended care wards at the intervention site
- Control Group- Post-Intervention: Medicine and extended care wards at control site
Arm/Group | Pre-Intervention Group | Control Group- Post-Intervention | Post-intervention Group
Number analyzed (Participants) | 169 | 65 | 157
Participants | 151 | 62 | 150

6. Secondary Outcome: Clinicians Acceptance of and Outcome Expectancy From Following the ABU Guidelines
Description: The investigators used a previous validated survey to measure this construct, which we termed "risk perception." We asked 5 questions, all exploring whether various patient characteristics (age, type of organism) might increase providers' sense that untreated ASB might be a risk to their patient's health. These questions were scored on a 1-5 scale, from strongly disagree to strongly agree, with 5 being the best answer (compliant with guidelines about ASB treatment), and 1 being the worst answer (least likely to comply with ASB guidelines). Higher scores mean a better answer. Lower scores mean a worse answer. The minimum value was 1, and the maximum value was 5. To create a score for this domain, we added up the score for each of the 5 questions and divided by the number of questions answered (by 5 if all 5 questions were answered; by 4 if only 4 of the 5 questions had been answered; etc).
Time Frame: one year
Population: health care practitioners
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group - Postintervention: Medicine and extended care wards at control site
Arm/Group | Pre-Intervention Group | Control Group - Postintervention | Post-intervention Group
Number analyzed (Participants) | 169 | 65 | 157
score on a scale | 3.0 (0.6) | 3.2 (0.5) | 3.3 (0.6)

7. Secondary Outcome: Number of Catheter-days of Use Per 1000 Patient Bed Days on Each Unit
Time Frame: One year
Population: inpatient-days on acute and extended care wards - aggregate numbers did not look at individual patients
Measure: Number; unit: catheter-days of use/1000 pt bed days
Units Other Than Participants: bed-days
Groups:
- Preintervention Acute Medical Care Line: Patients in acute medical care wards during the preintervention period
- Preintervention Extended Care Line: Patients in the extended care (nursing home) wards during the preintervention period
Arm/Group | Preintervention Acute Medical Care Line | Preintervention Extended Care Line
Number analyzed (Participants) | NA | NA
Number analyzed (bed-days) | 64699 | 63568
catheter-days of use/1000 pt bed days | 347.2 | 392.1

8. Secondary Outcome: Patient Level Analysis of Inappropriate Antibiotic Use
Description: The investigators looked at the percentage of cases of ASB (asymptomatic bacteriuria) that were inappropriately over-treated with antibiotics, and the percentage of cases of CAUTI (catheter-associated UTI) that were not treated with antibiotics (under-treated).
Time Frame: three years
Population: All patients on acute medical care wards or extended care wards during the three year study project who had a positive urine culture associated with the presence of a urinary catheter.
Measure: Number; unit: percentage of cases
Groups:
- Intervention Group: Cases of positive urine cultures on medicine and extended care wards at the intervention site
- Control Group: Cases of positive urine cultures on medicine and extended care wards at the control site
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 867 | 731
percentage of cases
  Year 1 ASB tx | 38 | 20
  Year 2 ASB tx | 22 | 25
  Year 3 ASB tx | 29 | 17
  Year 1 CAUTI not tx | 8 | 4
  Year 2 CAUTI not tx | 9 | 7
  Year 3 CAUTI not tx | 7 | 2
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.05, Regression, Logistic — We used χ2 test, Fisher's exact test and one-way ANOVA to determine if patient-level covariates differed between the baseline, intervention and maintenance periods at each study site

ADVERSE EVENTS:
Time Frame: All 3 years
Description: Only the under-treatment of CAUTI (failure to use antimicrobials when indicated) was collected/assessed/measured as an adverse event.
Arm/Group | Arm 1-Intervention: Audit-Feedback | Arm 2- Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 27/867 | 17/731
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Intervention: Audit-Feedback (N=867) | Arm 2- Control (N=731)
Incidence of under-treatment of CAUTI (Renal and urinary disorders) | 27 (27) | 17 (17)

LIMITATIONS AND CAVEATS:
Modification may be necessary for private sector facilities. We do not know what aspect of our intervention had the biggest impact, and whether the entire bundle is necessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes